CLINICAL TRIAL: NCT01466998
Title: Menopausal Treatment Using Relaxation Exercises (MaTURE)
Acronym: MaTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Deborah Grady, Professor of Medicine, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AT005491 (NIH)
Record Dates: First submitted 2011-11-01; First posted 2011-11-08 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Hot Flushes; Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paced Respiration (Experimental): Participants will use a small, commercially-available guided-breathing device to practice breathing at a rate slower than 10 breaths per minute. Participants will be instructed to use their devices for at least 15 minutes per day for 12 weeks.
  Interventions: Other: Paced Respiration
- Music Therapy (Active Comparator): Participant will use an identical appearing device, programmed to play quiet, relaxing non-rhythmic music while monitoring spontaneous breathing. Participants will be instructed to use their devices for at least 15 minutes per day for 12 weeks.
  Interventions: Other: Music Therapy

INTERVENTIONS:
Other: Paced Respiration — Practice paced respiration 15 minutes per day for a total of 12 weeks.
  Arms: Paced Respiration
Other: Music Therapy — Practice music therapy for 15 minutes per day for a total of 12 weeks.
  Arms: Music Therapy

SUMMARY:
Hot flashes occur in as many as two thirds of U.S. women during menopause and are severe enough to require treatment in 20%. Although postmenopausal hormone therapy is effective in suppressing hot flashes, it is associated with increased risk for a variety of serious adverse effects. There is an urgent need for alternative treatments that are effective, safe, and easy to use. In this study, the investigators will compare two different types of behavioral relaxation therapies, paced respiration and music therapy, for treatment of menopausal hot flashes. Effects on frequency of hot flashes, other symptom and quality-of-life outcomes associated with hot flashes, and physiologic measures of sympathetic/parasympathetic activity will be examined.

ELIGIBILITY:
Inclusion Criteria

1. Women aged 40 through 59 years at the time of screening.
2. Perinenopausal or postmenopausal.
3. Adequate adherence to study procedures during a 1-week run-in.
4. At least 4 hot flashes per 24 hours recorded by a hot flash monitor and diary.
5. Capable of understanding study procedures and giving informed consent.
6. Willing to refrain from using other treatments for hot flashes during the study period.

Exclusion criteria

1. Pregnant or breastfeeding in the past year.
2. Current or recent use of medications known to affect hot flashes.
3. Resting blood pressure less than 100/60.
4. Spontaneous resting breathing rate less than 10 breaths/minute.
5. Chronic medical therapy for pulmonary disease.
6. Known sensitivity to adhesives.
7. Cardiac pacemaker or implanted defibrillator.
8. No access to a telephone.
9. Plans to move out of the area or travel by airplane in ways that would interfere with the study.
10. Inability to sign an informed consent, participate in interviews, or understand and complete questionnaires in English.
11. Report conditions that, in the judgment of the investigators, render potential participants unlikely to follow the protocol.
12. Participation in another research study involving investigational drugs or devices.

Ages: 40 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in average daily frequency of hot flashes. | 4-Weeks and 12-Weeks

SECONDARY OUTCOMES:
Change in subjective severity of hot flashes. | 4-weeks and 12-weeks
Change in sympathetic and parasympathetic autonomic nervous system tone. | 12 weeks
Change in quality-of-of life measures associated with hot flashes. | Weeks 4 and Weeks 12

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Grady, MD, MPH, Principal Investigator — University of California, San Francisco; Alison Huang, MD, MAS, Study Director — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Huang AJ, Phillips S, Schembri M, Vittinghoff E, Grady D. Device-guided slow-paced respiration for menopausal hot flushes: a randomized controlled trial. Obstet Gynecol. 2015 May;125(5):1130-1138. doi: 10.1097/AOG.0000000000000821. PMID 25932840